CLINICAL TRIAL: NCT05515341
Title: A DirEct to PatieNt Study in Chronic Pain
Acronym: ENLITEN
Status: Recruiting | Type: Observational
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: A4102
Record Dates: First submitted 2022-08-23; First posted 2022-08-25 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Chronic Pain
Keywords: Chronic Pain
MeSH Terms: conditions — Chronic Pain | interventions — Therapeutics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Medical Device Therapy/Procedure for Chronic Pain
  Interventions: Device: Commercially Approved Interventional Medical Device/Therapy for Chronic Pain

INTERVENTIONS:
Device: Commercially Approved Interventional Medical Device/Therapy for Chronic Pain — Commercially Approved Interventional Medical Device/Therapy

SUMMARY:
To compile real-world, direct from patient clinical outcomes and objective metrics in patients who have received or plan to receive a commercially approved interventional medical device therapy/procedure for chronic pain in routine clinical practice.

ELIGIBILITY:
Key Inclusion Criteria:

* Patient is planning to receive or has received a commercially approved interventional medical device therapy/procedure to treat chronic pain, ascertained from self-reporting
* Age ≥ 22 years at time of eligibility screening, ascertained by self-reported age at time of eligibility screening
* Proficient in written and spoken English, defined by self-reporting of comfort reading, writing and speaking English

Key Exclusion Criteria:

* Requires a legal representative to sign the ICF ascertained from self-reporting

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Chronic pain
Sampling Method: Non-Probability Sample
Enrollment: 50000 (Estimated)
Dates: Start 2023-01-10 (Actual); Primary Completion 2029-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Change in pain post procedure | up to 12 months
  Change in patient-reported pain on a scale of 0 - 10 where 0 is no pain and 10 is maximum pain

CONTACTS AND LOCATIONS:
Overall Officials: Natalie B Lyons, Study Director — Boston Scientific Corporation
Locations (1):
- Boston Scientific Neuromodulation, Valencia, California, United States